CLINICAL TRIAL: NCT06042790
Title: Patients´ Mental and Physical Health After Being Treated for Covid-19 in an Intensive Care Unit in Sweden, a National Register Study
Brief Title: Patients´ Mental and Physical Health After Covid-19 Treated in ICU in Sweden
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Swedish Intensive Care Registry (Other)
Responsible Party: Principal Investigator, Sten Walther, Associate Professor, MD, Swedish Intensive Care Registry
Other Study IDs: SwedishICR
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Quality of Life; Intensive Care Unit Syndrome
Keywords: Covid 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid-19 ICU patients: Patients with confirmed Covid-19 admitted to ICU care
- non-Covid-19 patients: Non Coivd-19 patients admitted to ICU before 2020

SUMMARY:
Covid-19 is a disease where both clinical experience and thus knowledge about the long-term effects of the disease are currently sparse. However, current follow-up results indicate a more pronounced cognitive and respiratory impairment than previously seen in a normal ICU population. As we know that the prevalence of impairments in neurocognitive and Health Related Quality of Life (HRQoL) is increased in a majority of ICU patients, it would be of benefit to gain knowledge about the impact on the recovery trajectory for patients treated for Covid-19, and to increase the understanding of which factors that affect the HRQoL and recovery and in what way these differs between patients treated in ICU for Covid-19 and other causes respectively. This can contribute to better structures for follow-up and possibility to individualisation that better address which patients are in risk for decreased HRQoL and where benefit for the patient, health care and social economic can be achieved.

DETAILED DESCRIPTION:
Introduction During 2020, an infection disease caused by the new coronavirus Sars-Cov2, Covid-19 were globally spread in the world. Covid-19 caused extensive consequences to the society, economy, and health care. In some of the patients the symptoms progressed to a life-threatening respiratory failure whit a need for intensive care. The intensive care was complicated then the progress of the disease was not followed the usual care for patients with difficult respiratory disease. Many of the patients with Covid-19 required deeper sedation with high-doses of anaesthesia and muscle relaxants and long time in ventilator. This is not in line with the current evidence regarding ventilator treatment and sedation in intensive care and for considered to constitute risk-factors for intensive care related residuals symptoms and worsened long-time results as well as increased mortality. In addition, the hospitals had restrictions regarding visitors and the relatives were not allowed to visit patients at the Intensive Care Unit (ICU). The presence of relatives is estimated in intensive care patients as one of the most important factors contributing to their recovery.

Today we know that intensive care patients had a risk to get physical, mental, and cognitive problems long time after hospital discharge. Other common residual problems as anxiety, depression, and post-traumatic stress (PTSD) can also occurred after intensive care. However, there are an increased risk that ICU patients with Covid-19 experience physical, and mental problems and decreased health related quality of life (HRQoL), then the environment at ICU during the Covid-19 pandemic, could predispose for cognitive failure and PTSD. The knowledge about this is limited. Today, data indicate that fatigue and dyspnoea are common residual symptoms which affect the HRQoL in multiple dimensions long time after hospital discharge.

Since 2005 the Swedish Intensive Care Registry (SIR) recommend to follow-up former ICU patients HRQoL (RAND-36), BMI, ADL and working capacity. We have now a unique chance to describe how patients taken care for Covid-19 in ICU experience their HRQoL with physical, mental, and cognitive problems compared to patients who were cared for in ICU for reasons other than Covid-19, and if they changed over time in relation to changed treatment conditions. It is important to map which risk factors that affect patients HRQoL. International studies show that factors important to HRQoL after intensive care are: age, comorbidity, the severity of the illness, length of stay, diagnose, PTSD, and symptoms of depression. It is likely that other factors also play a decisive role, such as socioeconomics factors. The purpose of this study is to deepen the analyse and identify other factors that are important for the patients HRQoL.

Aim The aim is to increase the knowledge about adult patient's whit Covid-19 taken care of at ICUs in Sweden estimate their HRQoL during the first year after ICU discharge and compare their HRQoL with patients taken care at ICU for other reasons than Covid-19 and which risk-factors affect the HRQoL and if there are any discrepancy between the groups.

Research-questions Are there differences in self-estimated HRQoL between patients care for Covid-19 and patients cared for other reasons at ICU, at 3, 6 and 12 months after ICU discharge? Method Design: National quality register study. Participants/sample size: All adult patients ≥18 year who have been treated at ICUs in Sweden and have a registered follow-up in SIR. (Covid-19 and non-Covid-19).

Data Collection:

Anonymous data collected from the Swedish intensive quality register (SIR), the national patient register in the National board of health and welfare, and the Statistics Sweden (SBC) LISA register for patients cared for in ICU and how have a registered RAND-36 in SIR. The Covid-19 group include patients cared in ICU between 01-03-2020 and as long as the pandemic is ongoing. The non-Covid-19 group includes patients how have been cared in ICU 01-01-2017 until 31-12-2019, before the outbreak of the pandemic to get the best comparing data. The reasons to include data from SIR are 1) to reduce the effort for the patients, to fill in more questionnaires and 2) that the time before outbreak of Covid-19 is more valid to compare with then the intensive care during the Covid-19 pandemic have to deviate from their usual regimen regarding care and treatment as well as the selection of patients and a comparison during the Covid period therefore has a risk of bias Data analysis Data compiled on group-level and to be used to compare between the groups. Quantitative methods are used to describe tendances in the group and analysis of differences between the groups. Data regarding demography and comorbidity analysis descriptively at group level.

Association is investigated with correlation and regression analysis, t-test or corresponding.

Comparison between the groups is done with t-test parametric data and Mann-Whitney non-parametric variables. Identifying of factors influencing the outcome of RAND-36 (HRQoL) is done with univariate regression analysis. Values with significant outcomes are further analysed with multivariate regression analysis for identification of independent risk factors versus outcomes in RAND-36 (HRQoL). The results of variate analysis reports as OR.

ELIGIBILITY:
Inclusion Criteria:

Consecutively admitted ICU patients with a completed RAND-36 follow-up form

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group I ICU patients with Covid-19 Group II ICU patients without Covid-19
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2023-10-08 (Estimated)

PRIMARY OUTCOMES:
HRQoL | 2, 6, 12 months post ICU
  RAND-36

CONTACTS AND LOCATIONS:
Overall Officials: Sten Walther, PhD, Study Chair — Linkoeping University
Locations (1):
- The Swedish Intensive Care Registry, Karlstad, Sweden

IPD SHARING:
Plan to Share IPD: No